CLINICAL TRIAL: NCT02881593
Title: Study of the Quality of the Release on Postoperative Scanners in Minimally Invasive Arthrodesis
Brief Title: Study of the Quality of Post Release on Scanners Operating in Minimally Invasive Arthrodesis
Status: Withdrawn | Type: Observational
Why Stopped: The investiagtor abandoned the project.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ARTHROSCAN
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Arthrodesis
Keywords: Operating in Minimally Invasive
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
For twenty years, as for other surgical disciplines, new minimally invasive techniques have been developed with the main goal the reduction of muscle trauma associated with the surrounding roads "classic" and reduce morbidity linked to this one.

More recently, minimally invasive methods dedicated to spinal surgery were established, for the treatment of herniated discs initially, then for narrow lumbar canals.

The canal release on minimally invasive fusion, using a tubular system for muscle retraction is a new technique that has proven effective: post operative pain reduction of hospital stay and blood loss.

The objective of the study is to investigate the quality of ductal release in these minimally invasive fusions.

Main objective of the study: Evaluation of the quality of the release of post scanners operative minimally invasive arthrodesis

Secondary Objectives: Assessment rates/types of early complications of technical Minimally invasive - early postoperative results (postoperative pain, analgesic consumption, length of hospital stay, blood loss) - in clinical outcomes in the short and medium term decompression after minimally invasive fusion.

DETAILED DESCRIPTION:
I. Background / Rationale

For twenty years, as for other surgical disciplines, new minimally invasive techniques have been developed with the main goal the reduction of muscle trauma associated with the surrounding roads "classic" and reduce morbidity linked to this one.

More recently, minimally invasive methods dedicated to spinal surgery were established, for the treatment of herniated discs initially, then for narrow lumbar canals.

The canal release on minimally invasive fusion, using a tubular system for muscle retraction is a new technique that has proven effective: post operative pain reduction of hospital stay and blood loss.

The objective of the study is to investigate the quality of ductal release in these minimally invasive fusions.

II. objectives

at. primary objective

Evaluating the quality of discharge on postoperative scanners minimally invasive fusions.

b. secondary objectives

i. Evaluation of the rate and type of early complications in the minimally invasive technique

ii. Evaluation of early postoperative results (postoperative pain, analgesic consumption, length of hospital stay, blood loss)

iii. Evaluation of clinical outcomes in the short and medium term decompression after minimally invasive fusion.

III. Methodology and duration of the research

This is a retrospective single-center consecutive series multi-operator regarding the evaluation of surgical practice cited in goal.

Clinical data were collected prospectively by KEOPS database (SAMIO). All patients included in our study have spinal MRI scanners and pre-operative and post-operative scans.

N = (number of patients and over what period) / Time Study?

The series of patients will be classified into two groups:

* Foraminal stenosis
* Central stenosis

The evaluation of the primary objective criterion is comparing the height of the foramen measured on CT pre- and post-operative between the lower edge of the overlying pedicle and the top edge of the pedicle underlying the sagittal sections.

For central stenosis, Postoperative MRI will be performed and the volume of the dural sac will be compared to preoperative MRI on axial images.

ELIGIBILITY:
Inclusion Criteria:

* Ductal compression on one floor
* Scanner spine preoperatively

Exclusion Criteria:

* Spondylolisthesis significant (greater than grade 2)
* Stenoses multi layered
* Major spinal deformities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with Paris Saint Joseph with canal compression on one floor, for whom a scan of the spine is performed preoperatively
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02-02 (Estimated); Primary Completion 2015-02-02 (Estimated); Study Completion 2015-02-02 (Estimated)

PRIMARY OUTCOMES:
comparing the measured height of the foramen on the CT scanner | Day -1 and Day 1 after surgery
  The evaluation of the primary objective criterion is comparing the height of the foramen measured on CT pre- and post-opéraoires between the lower edge of the overlying pedicle and the top edge of the pedicle underlying the sagittal sections.
Assessment of change of MRI volume of dural sac | Day -1 and Day 1 after surgery
  For central stenosis, Postoperative MRI will be performed and the volume of the dural sac will be compared to preoperative MRI on axial slices

SECONDARY OUTCOMES:
Assessment of change of Oswestry score | Day -1 and Day 1 after surgery
  Oswestry score (<30%: State almost normal 30 to 50%: Moderate disability 50% to 70%: Severe disability> 70%: full disability)
Evaluation of pain by visual analogue scale VAS | Day -1 and Day 1 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume P RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph

IPD SHARING:
Plan to Share IPD: Undecided